CLINICAL TRIAL: NCT04720833
Title: Effect of Dried Plum on Bone and Markers of Bone Status in Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Shirin Hooshmand, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2521098
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Prunes; dried plum; nutrition; bone
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Calcium; Vitamin D

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assign to one of the arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dried plum (100 g dried plum) (Experimental): Participants will receive 100 g dried plum daily plus 500 mg calcium and 300 IU vitamin D daily
  Interventions: Dietary Supplement: dried plum
- Calcium and vitamin D (Placebo Comparator): Participants will receive 500 mg calcium and 300 IU vitamin D daily
  Interventions: Dietary Supplement: Calcium and vitamin D

INTERVENTIONS:
Dietary Supplement: dried plum — Dried plum
  Arms: dried plum (100 g dried plum)
Dietary Supplement: Calcium and vitamin D — Calcium and vitamin D supplement
  Arms: Calcium and vitamin D

SUMMARY:
The principal objective of this study is to examine whether the addition of 100 g dried plum to the diets of men, regardless of their bone status, positively influences their indices of bone turnover in comparison with their corresponding baseline values and the control regimen.

DETAILED DESCRIPTION:
To test the bone protective properties of dried plum, 66 men (50 to 79 years of age) will receive either 100 g dried plum/day or a control regimen for 12 months. Both groups will receive 500 mg calcium and 400 IU vitamin D daily.

Evaluation will be based on analyses of bone mineral density at baseline, 6 and 12-months and serum and urine markers of bone formation and resorption at baseline and 3, 6, and 12-months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men (50-79 year-old)

Exclusion Criteria:

* endocrine (e.g., prednisone, other glucocorticoids) or neuroactive (e.g., dilantin, phenobarbital) drugs or any drugs known to influence bone and calcium metabolism
* Men whose BMD t-score at any site falls below 2.5 SD of the mean will be excluded from the study and referred to their primary care physician
* subjects treated with calcitonin, bisphosphonates, raloxifene, sodium fluoride, anabolic agents, e.g. PTH and growth hormone, or steroids for less than 3 months prior to the start of the study will be excluded.
* body mass index (BMI) <18 and >30 will be excluded to avoid extremes in leanness/adiposity and to readily allow body composition assessment.
* If subjects smoke 20 cigarettes or more per day, they will be excluded.
* Men who regularly consume dried plum or prune juice will not be accepted into the study.

Ages: 50 Years to 79 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Bone biomarkers | changes from baseline to 3 months
  TRAP5b, BAP, CTX, P1NP

SECONDARY OUTCOMES:
Bone mineral density | changes from baseline to 12 months
  BMD by DXA

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Hooshmand, PhD, RD, Principal Investigator — San Diego State University
Locations (1):
- School of Exercise and Nutritional Sciences, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hooshmand S, Gaffen D, Eisner A, Fajardo J, Payton M, Kern M. Effects of 12 Months Consumption of 100 g Dried Plum (Prunes) on Bone Biomarkers, Density, and Strength in Men. J Med Food. 2022 Jan;25(1):40-47. doi: 10.1089/jmf.2021.0080. Epub 2021 Oct 29. PMID 34714130